CLINICAL TRIAL: NCT00189969
Title: Phase I Study to Evaluate Take Rate, Immunogenicity and Safety of Bavarian Nordic's Smallpox Vaccine Elstree-BN Administered to Healthy Vaccinia-Naive Subjects in the Age of 18-32 Years
Brief Title: Take Rate, Immunogenicity and Safety of Elstree-BN Smallpox Vaccine in Healthy Vaccinia-Naive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: POX-ELS-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-04-21 (Estimated); Status verified 2006-04

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox

INTERVENTIONS:
Biological: Elstree-BN

SUMMARY:
The purpose of this study is to assess the take rate (formation of a typical postvaccinal lesion)and the safety and immunogenicity of the smallpox vaccine Elstree-BN.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Free of obvious health problems
* Negative HIV test
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus
* Hematocrit ≥ 38%; white blood cells between 4.0 and 10.0 / nl with differential blood count without clinical finding; and platelets between 150 and 400 / nl
* ALT < 1.5 times institutional upper limit of normal
* Negative urine glucose by dipstick or urinalysis
* Adequate renal function defined as a serum creatinine < 1.5 mg/dL; urine protein < 100 mg/dL or < 2+ proteinuria; and a calculated creatinine clearance > 55 mL/min.
* For women, negative pregnancy test at screening and within 24 hours prior to vaccination.
* If the volunteer is female and of childbearing potential, she agrees to use acceptable contraception.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Known or suspected history of smallpox vaccination
* Typical vaccinia scar
* Vaccinia specific antibodies at screening
* History of immunodeficiency
* Known or suspected impairment of immunologic function
* Use of immunosuppressive medication or radiation therapy
* Any history of atopic disease
* Eczema of any degree or history of eczema
* Chronic exfoliative skin disorders/conditions or any acute skin disorders of large magnitude
* Any malignancy including leukemia or lymphoma
* Presence of any infectious disease or a history or evidence of autoimmune disease
* History or clinical manifestation of clinically significant mental illness or haematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders
* History of drug or chemical abuse
* Administration of inactivated vaccine 14 days prior to vaccination
* Any immune modifying therapy within 4 weeks prior to vaccination
* Administration of live attenuated vaccines within 60 days prior to vaccination
* Receipt of blood products or immunoglobulin in the past 6 months
* Subjects with acute febrile illness within one week prior to vaccination or subjects who may be in the incubation period of an infectious disease
* Household contacts/sexual contacts with, or occupational exposure to any of the following:

  1. Pregnant women
  2. Children <12 months of age
  3. People with current or history of atopic dermatitis
  4. People with chronic exfoliative skin disorders/conditions or any acute skin disorders
  5. People with immunodeficiency disease, malignancies or use of immunosuppressive medications
* History of anaphylaxis or severe allergic reaction
* Hypersensitivity to egg or chick protein
* Known allergies to any component of the vaccine or its diluent
* Known allergies to any known component of VIG
* Known allergies to cidofovir or probenecid
* Abnormalities suggestive of any underlying disease, detected at routine tests prior to study inclusion
* Use of any investigational or non-registered drug or vaccine starting 30 days preceding the study vaccine and ending at conclusion visit
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor.
* Three or more of the following risk factors: An immediate family member who has had onset of ischemic heart disease before age 50 years, elevated blood pressure, elevated blood cholesterol, diabetes or nicotine abuse.

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2003-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Occurrence of a typical pock ("take") which is associated historically with protection against variola within one week after vaccination.

SECONDARY OUTCOMES:
Occurrence, relationship and intensity of any serious adverse event at any time during the study / any non-serious adverse event within 4 weeks after vaccination.
ELISA / Neutralisation assay specific seroconversion rates and geometric mean titres 2,4,12,52 and 104 weeks after vaccination.
Interferone-gamma producing T cells 2,4,12,52 and 104 weeks after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Schroedter, M.D., Principal Investigator — Focus Clinical Drug Development GmbH
Locations (1):
- Focus Clinical Drug Development GmbH, Neuss, Nordrhein, Germany